CLINICAL TRIAL: NCT00272896
Title: Hemodynamic and Headache-Inducing Effect of Intravenous Vasoactive Intestinal Peptide (VIP) in Migraineurs
Brief Title: Hemodynamic and Headache-Inducing Effect of Intravenous Vasoactive Intestinal Peptide in Migraineurs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danish Headache Center (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: KA04119
Record Dates: First submitted 2006-01-04; First posted 2006-01-09 (Estimated); Last update posted 2006-01-09 (Estimated); Status verified 2004-10

CONDITIONS: Headache; Migraine; Vasoactive Intestinal Peptide; Ultrasonography, Doppler, Transcranial
Keywords: Migraine; VIP; Transcranial Doppler; Headache
MeSH Terms: conditions — Headache; Migraine Disorders | interventions — Vasoactive Intestinal Peptide

INTERVENTIONS:
Drug: Vasoactive intestinal peptide

SUMMARY:
We hypothesized that infusion of VIP may induce headache/migraine in migraineurs and that VIP-induced headache may be associated with dilation of intra- and extracranial vessels. To test this hypothesis, we performed a double blind placebo-controlled crossover study in migraineurs and studied the effect on headache and cerebral and systemic hemodynamic parameters.

DETAILED DESCRIPTION:
We hypothesized that infusion of VIP may induce headache/migraine in migraineurs and that VIP-induced headache may be associated with dilation of intra- and extracranial vessels. To test this hypothesis, we performed a double blind placebo-controlled crossover study in migraineurs and studied the effect on headache and cerebral and systemic hemodynamic parameters. The subjects were randomly allocated to the infusion of 8pmol/kg/min VIP or placebo (isotonic saline), duration 25min. Headache intensity, mean velocity of blood flow in the middle cerebral artery (VmMCA), superficial temporal artery diameter, end-expiratory CO2 and vital signs were recorded at baseline and then every 10 min until 120 min after start of the infusion. The patients received a headache diary for the following 12 hours after infusion.

ELIGIBILITY:
Inclusion Criteria:

* migraineurs

Exclusion Criteria:

* cerebrovascular disorders, pregnancy, nursing

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12
Dates: Start 2004-10; Study Completion 2005-09

PRIMARY OUTCOMES:
Headache
Intra- and extracranial vasodilation

SECONDARY OUTCOMES:
arterial blood pressure
heart rate

CONTACTS AND LOCATIONS:
Overall Officials: Jes Olesen, MD, PhD, Principal Investigator — Danish Headache Center, Glostrup, Denmark
Locations (1):
- Glostrup Hospital, Glostrup Municipality, Denmark